CLINICAL TRIAL: NCT01005381
Title: The Effect of Particle Size of Calcium Carbonate and Vitamin D on Calcium and Bone Parameters in Adolescent Girls
Brief Title: Effect of Calcium Supplement Particle Size and Vitamin D Supplement on Calcium Retention in Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 0609004386
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis
Keywords: Calcium; Vitamin D; Particle Size; Adolescents; Bone; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Small Particle Size Calcium Carbonate (Experimental): Subjects are given small particle size calcium carbonate supplement twice daily (total of 625 mg/d from supplement).
  Interventions: Dietary Supplement: Small Particle Size Calcium Carbonate Supplement
- Large Particle Size Calcium Carbonate (Active Comparator): Subjects are given a large particle size calcium carbonate supplement twice daily (total of 625 mg/d from supplement).
  Interventions: Dietary Supplement: Large Particle Size Calcium Carbonate Supplement
- Calcium Placebo (Placebo Comparator): Subjects are given two placebo tablets daily, which are identical to the large and small particle size calcium carbonate supplements.
  Interventions: Dietary Supplement: Calcium Placebo
- No Vitamin D supplement (Active Comparator): Subjects are given calcium carbonate supplement once daily (325 mg/d from supplement).
  Interventions: Dietary Supplement: Small Particle Size Calcium Carbonate Supplement
- Vitamin D supplement (Experimental): Subjects are given a calcium supplement once daily (325 mg/d from supplement) with 1000 IU/d vitamin D supplement.
  Interventions: Dietary Supplement: Small Particle Size Calcium Carbonate Supplement; Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Small Particle Size Calcium Carbonate Supplement — Small Particle Size Calcium Carbonate - tablet, 325 mg/tablet. Given once or twice daily depending on study arm.
  Arms: No Vitamin D supplement; Small Particle Size Calcium Carbonate; Vitamin D supplement
Dietary Supplement: Large Particle Size Calcium Carbonate Supplement — Large Particle Size Calcium Carbonate Supplement - tablet, 325 mg/tablet. Given twice daily.
  Arms: Large Particle Size Calcium Carbonate
Dietary Supplement: Vitamin D — Vitamin D - capsule, cholecalciferol, 1000 IU/tablet. Given once daily.
  Arms: Vitamin D supplement
Dietary Supplement: Calcium Placebo — Placebo tablets identical to the large and small particle size calcium carbonate tablets.
  Given twice daily.
  Arms: Calcium Placebo

SUMMARY:
This study has two research arms:

The purpose of the 1st is to determine if a smaller particle size calcium carbonate supplement (than that which is now commercially available) improves calcium absorption and retention in adolescents girls.

The purpose of the 2nd is to determine if vitamin D supplementation improves calcium absorption and retention in adolescents girls.

DETAILED DESCRIPTION:
An important strategy to reducing the risk for osteoporosis and fracture in later life is to optimize the development of peak bone mass during adolescence. Because calcium is the main mineral component of bone, maximizing calcium absorption and retention during adolescence is important to maximize peak bone mass.

Our two research arms address two different mechanisms by which calcium absorption and retention may be increased:

1. We hypothesize that a smaller particle size calcium carbonate supplement (than that which is now commercially available) may be better absorbed and lead to higher calcium retention in adolescents.
2. We hypothesize that vitamin D supplementation will increased calcium absorption and retention in adolescents.

Subjects will be assigned to one of the two research arms.

1)Small and large particle size calcium supplements or placebo or 2) calcium supplements with or without vitamin D supplements will be given to subjects during two 3-week study periods in which subjects live on-site.

Calcium absorption will be measured by parathyroid hormone suppression after a calcium load and by stable calcium isotope in some subjects.

Calcium retention will be measured by calcium intake minus calcium excretion.

ELIGIBILITY:
Inclusion Criteria:

* 12-14 year old girls
* Generally Healthy

Exclusion Criteria:

* History of alcohol, smoking, or non-prescription drug use
* Malabsorptive disorders, bone, liver, or kidney disease that may affect calcium metabolism
* Oral contraceptive use
* Pregnancy

Ages: 12 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Calcium Balance | weeks 2,3 + 5,6
  Total calcium(Ca) retention will be calculated - Ca retention/d = Ca intake/d - Ca excretion/d (urine + feces)
Calcium Absorption | Day 15, 30

SECONDARY OUTCOMES:
Serum parathyroid hormone suppression | Day 19, 40
  Serum PTH will be measured by a 2-site immunoassay
Serum 25-hydroxyvitamin D | Day 1, 20, 2, 41
  Serum 25-hydroxyvitamin Dwill be measured by LCMS
Urinary Calcium | Weeks 2,3 + 5,6
  Ca content of all 24 h urine collections will be measured by Atomic Absorption Spectrophotometry
Fecal Calcium | Weeks 2,3 + 5,6
  Ca content of all fecal collections will be measured by Atomic Absorption Spectrophotometry

CONTACTS AND LOCATIONS:
Overall Officials: Connie M Weaver, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Park CY, Hill KM, Elble AE, Martin BR, DiMeglio LA, Peacock M, McCabe GP, Weaver CM. Daily supplementation with 25 mug cholecalciferol does not increase calcium absorption or skeletal retention in adolescent girls with low serum 25-hydroxyvitamin D. J Nutr. 2010 Dec;140(12):2139-44. doi: 10.3945/jn.110.124891. Epub 2010 Oct 20. PMID 20962148